CLINICAL TRIAL: NCT00300521
Title: Liver Transplantation With ADV-TK Gene Therapy Improves Survival in Patients With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Collaborators: Tongji University (Other); The No.180 Hospital of People's Liberation Army (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LT2000-09
Record Dates: First submitted 2006-03-08; First posted 2006-03-09 (Estimated); Last update posted 2006-03-09 (Estimated); Status verified 2000-09

CONDITIONS: Hepatocellular Carcinoma; Liver Transplantation
Keywords: hepatocellular carcinoma; liver transplantation; adenovirus-thymidine kinase enzyme; gene therapy; immunosuppression
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Genetic Therapy

INTERVENTIONS:
Genetic: ADV-TK (adenovirus-thymidine kinase enzyme) gene therapy

SUMMARY:
Previous rather poor results in liver transplantation (LT) of patients with advanced hepatocellular carcinoma (HCC) have made the application of LT very limited in treatment of HCC. The advantages of ADV-TK gene therapy highlight its potentiality as adjuvant treatment for HCC patients after LT. We reported here the improved outcome of LT with combined treatment of ADV-TK gene therapy in patients with intermediate or advanced HCC.

DETAILED DESCRIPTION:
The overall survival in the LT with ADV-TK gene therapy group was 54.8 % at three years, and the recurrence-free survival in the same group was 56.5 %, both being higher than those in the transplantation only group (P=0.0001 for overall survival and P=0.0000 for recurrence-free survival). In no-vascular invasion subgroup treated with LT with ADV-TK therapy, both overall survival and recurrence-free survival were 100 %, significantly higher than those with vascular invasion subgroup treated with the combined LT and ADV-TK therapy (P=0 for each group). Vascular invasion was an important factor affected survival and recurrence, hazard ratio=3.687; P=0.014 and hazard ratio=12.961; P=0.000, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of advanced hepatocellular carcinoma with no metastasis in lungs and bones
* Accept Liver Transplantation

Exclusion Criteria:

* Small hepatocellular carcinoma
* Advanced hepatocellular with metastasis in lungs and bones

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2000-09; Study Completion 2005-11

PRIMARY OUTCOMES:
overall survival rate at one year
overall survival rate at two year
overall survival rate at three year
overall recurrence-free survival rate at one year
overall recurrence-free survival rate at two year
overall recurrence-free survival rate at three year

SECONDARY OUTCOMES:
AFP level before and after liver transplantation
hazard rate of age on survival rate and recurrence-free survival rate
hazard rate of TNM stage on survival rate and recurrence-free survival rate
hazard rate of Child-Pugh classification on survival rate and recurrence-free survival rate
hazard rate of vascular invasion on survival rate and recurrence-free survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Ding Ma, M.D., Study Chair — Cancer Biology Research Center, Tongji Hospital, Tongji Medical college, Huazhong University of Science and Technology, Wuhan, Hubei 430030, P.R.China; Ning Li, B.D, Study Director — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chao Yang Hospital, Beijing, Beijing Municipality, China